CLINICAL TRIAL: NCT03198026
Title: Phase II, Single Arm, Open Label Multi-center Study of Obinutuzumab and Ibrutinib in the Front Line Treatment of Indolent Non-Hodgkin's Lymphomas
Brief Title: Obinutuzumab and Ibrutinib as Front Line Therapy in Treating Patients With Indolent Non-Hodgkin's Lymphomas
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Sidney Kimmel Cancer Center at Thomas Jefferson University (Other)
Collaborators: Genentech, Inc. (Industry); Pharmacyclics LLC. (Industry)
Responsible Party: Sponsor
Organization: Thomas Jefferson University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 17P.176; JT 10049 (Other: JeffTrial Number)
Record Dates: First submitted 2017-06-22; First posted 2017-06-23 (Actual); Last update posted 2025-08-22 (Actual); Status verified 2025-08

CONDITIONS: Non-Hodgkin's Lymphoma; Ann Arbor Stage II Extranodal Marginal Zone Lymphoma of Mucosa-Associated Lymphoid Tissue; Ann Arbor Stage II Follicular Lymphoma; Ann Arbor Stage II Nodal Marginal Zone Lymphoma; Ann Abor Stage III B-Cell Non-Hodgkin Lymphoma; Ann Arbor Stage III Extranodal Marginal Zone Lymphoma of Mucosa-Associated Lymphoid Tissue; Ann Arbor Stage III Follicular Lymphoma; Ann Arbor Stage III Nodal Marginal Zone Lymphoma; Ann Arbor Stage IV B-Cell Non-Hodgkin Lymphoma; Ann Arbor Stage IV Extranodal Marginal Zone Lymphoma of Mucosa-Associated Lymphoid Tissue; Ann Arbor Stage IV Follicular Lymphoma; Ann Arbor Stage IV Nodal Marginal Zone Lymphoma; Grade 1 Follicular Lymphoma; Grade 2 Follicular Lymphoma; Grade 3a Follicular Lymphoma; Indolent Non-hodgkin Lymphoma; Stage II Splenic Marginal Zone Lymphoma; Stage III Splenic Marginal Zone Lymphoma; Stage IV Splenic Marginal Zone Lymphoma
MeSH Terms: conditions — Lymphoma, Non-Hodgkin; Lymphoma, Follicular | interventions — ibrutinib; obinutuzumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (ibrutinib, obinutuzumab) (Experimental): Patients receive ibrutinib orally (PO) once daily (QD) on days 1-28. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity. Patients also receive obinutuzumab intravenously (IV) on days 1, 8, and 15 of cycle 1 and day 1 of subsequent cycles. Treatment repeats every 28 days for up to 6 cycles in the absence of disease progression or unacceptable toxicity. Beginning 2 months after cycle 6, patients with stable disease will continue to receive obinutuzumab every 2 months for a total of 12 doses.
  After completion of study treatment, patients are followed up monthly for 1 year, every 3-6 months for 4 years, and then annually for up to 2 years.
  Interventions: Drug: Ibrutinib; Biological: Obinutuzumab; Other: Laboratory Biomarker Analysis

INTERVENTIONS:
Drug: Ibrutinib — Given PO
  Other Names: 2-Propen-1-one; 1-((3R)-3-(4-amino-3-(4-phenoxyphenyl)-1h-pyrazolo(3,4-d)pyrimidin-1-yl)-1-piperidinyl)-; BTK Inhibitor PCI-32765; CRA-032765; Imbruvica; PCI-32765; 936563-96-1
Biological: Obinutuzumab — Given IV
  Other Names: 949142-50-1; Anti-CD20 Monoclonal Antibody R7159; Gazyva; R7159; RO 5072759; GA-101; GA101; huMAB(CD20); RO-5072759; RO5072759
Other: Laboratory Biomarker Analysis — Correlative studies

SUMMARY:
This phase II trial studies how well obinutuzumab and ibrutinib work as front line therapy in treating patients with indolent non-Hodgkin's lymphoma. Monoclonal antibodies, such as obinutuzumab, may interfere with the ability of cancer cells to grow and spread. Ibrutinib may stop the growth of cancer cells by blocking some of the enzymes needed for cell growth. Giving obinutuzumab and ibrutinib may work better in treating patients with non-Hodgkin's lymphomas.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To assess the efficacy of the combination of ibrutinib and obinutuzumab in chemotherapy naive patients with indolent lymphomas.

SECONDARY OBJECTIVES:

I. To assess progression free survival rates and overall survival rates in indolent lymphomas.

II. To assess safety and tolerability of the combination. III. To evaluate response using positron emission tomography (PET) and correlate PET negativity with durability of response.

OUTLINE:

Patients receive ibrutinib orally (PO) once daily (QD) on days 1-28. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity. Patients also receive obinutuzumab intravenously (IV) on days 1, 8, and 15 of cycle 1 and day 1 of subsequent cycles. Treatment repeats every 28 days for up to 6 cycles in the absence of disease progression or unacceptable toxicity. Beginning 2 months after cycle 6, patients with stable disease will continue to receive obinutuzumab every 2 months for a total of 12 doses.

After completion of study treatment, patients are followed up monthly for 1 year, every 3-6 months for 4 years, and then 1 year later.

ELIGIBILITY:
Inclusion Criteria:

* Previously untreated, histologically confirmed indolent non-Hodgkin's lymphoma as follows:

  * Follicular lymphoma (World Health Organization [WHO] classification grade 1, 2, or 3a)
  * Marginal zone lymphoma including:

    * Nodal and splenic marginal zone lymphoma (MZL) who have an indication for systemic therapy
    * Extranodal MZL:

      * Nongastric/noncutaneous MZL requiring systemic therapy
      * Cutaneous MZL will be eligible only if they have pathologically confirmed extra-cutaneous disease
      * Gastric MZL only if stage IIIE/IV defined as lymph node involvement on both sides of the diaphragm or with disseminated extranodal disease such as bone marrow or additional extra nodal sites
* Pathological diagnosis should be obtained by incisional or excisional tissue biopsy; core biopsy is permissible if obtaining an incisional or excisional is not possible and if the grade can be assessed on the core biopsy; a core biopsy can also be used if deemed in the best interest of the patient in the opinion of the investigator
* Patients must have stage II-IV disease
* All patients should have measurable disease; measurable disease is defined as a lymph node or tumor mass that is >= 1.5 cm in at least one dimension by computed tomography (CT) or the CT portion of the PET/CT
* Documentation of CD20+ status
* Patients must have an indication for therapy per standard modified Groupe d'Etude des Lymphomes Folliculaires (GELF) criteria including:

  * Symptoms attributable to lymphoma
  * B symptoms
  * Threatened end-organ function
  * Pleural effusions or peritoneal ascites
  * Cytopenia secondary to lymphoma
  * Leukemia
  * Bulky disease (defined as: Single mass >7cm in diameter, or 3 or more masses > 3 cm in diameter)
  * Splenomegaly
  * And steady progression over at least 6 months
* Age > 18 years
* Eastern Cooperative Oncology Group (ECOG) performance status 0-2
* Patients must be able to swallow whole pills
* Ability and willingness to comply with the requirements of the study protocol; when it is determined by the study investigator that a potential research participant is cognitively impaired, a surrogate consent from a caregiver or legally-authorized representative will be obtained. Caregiver or legally-authorized representative will ensure that they comply with the protocol in order for the subject to be considered eligible
* Female subjects who are of non-reproductive potential (i.e., post-menopausal by history - no menses for >= 1 year; OR history of hysterectomy; OR history of bilateral tubal ligation; OR history of bilateral oophorectomy); female subjects of childbearing potential must have a negative urine/serum pregnancy test upon study entry
* Male and female subjects who agree to use both a highly effective method of birth control (e.g., implants, injectables, combined oral contraceptives, some intrauterine devices [IUDs], complete abstinence , or sterilized partner) and a barrier method (e.g., condoms, vaginal ring, sponge, etc) during the period of therapy; female patients of reproductive potential who are not surgically sterile must practice adequate birth control for a minimum of twelve months post-treatment; male patients who are not surgically sterile must practice adequate birth control for a minimum of three months post-treatment
* Absolute neutrophil count > 1.5 x 10^9 cells/mm^3
* Platelet count > 50,000 cells/mm^3 (50 x 10^9/L)
* Hemoglobin > 9.0 g/dL
* Serum aspartate transaminase or alanine transaminase =< 3.0 x upper limit of normal (ULN)
* Prothrombin time (PT)/international normalized ratio (INR) < 1.5 x ULN and activated partial thromboplastin time (aPTT) < 1.5 x ULN (unless abnormalities are unrelated to coagulopathy or bleeding disorder)
* Estimated creatinine clearance >= 30 ml/min (calculated according using Cockcroft-Gault formula)
* Bilirubin =< 1.5 x ULN (unless bilirubin rise is due to Gilbert's syndrome or of non-hepatic origin)
* Patients with Child Pugh B or C liver failure will be excluded

Exclusion Criteria:

* Prior history of malignancies unless the patient has been disease free for >= 5 years; exceptions include basal cell carcinoma or squamous cell carcinoma of the skin; carcinoma in situ of cervix; carcinoma in situ of breast, localized prostate cancer, or superficial bladder cancer that has undergone curative therapy
* Prior therapy for lymphoma including chemotherapy or immunotherapy including ibrutinib/anti-CD20 agents; patient may have received corticosteroids, but should be off them 2 weeks prior to study entry; known prior significant hypersensitivity to obinutuzumab (not including infusion reactions) or ibrutinib
* Patients with evidence of large B cell transformation (transformed disease) are not eligible
* Known central nervous system (CNS) involvement by lymphoma
* Known bleeding disorders (e.g., von Willebrand's disease or hemophilia)
* Concomitant use of warfarin or other vitamin K antagonists
* Requires treatment with a strong cytochrome P450 (CYP) 3A inhibitor
* Known active bacterial, viral, fungal, mycobacterial, or other infection (excluding fungal infections of nail beds) or any major episode of infection requiring treatment with IV antibiotics or hospitalization (related to the completion of the course of antibiotics) within 4 weeks before the start of cycle 1
* Known infection with human immunodeficiency virus (HIV) or human T-cell leukemia virus 1 (HTLV-1) seropositive status
* Viral hepatitis:

  * Patients with active hepatitis B defined by hepatitis B surface antigen positivity or core antibody positivity in the presence of detectable serum hepatitis B deoxyribonucleic acid (DNA) viremia are not eligible for this study
  * Patients with a positive hepatitis B core antibody but with negative hepatitis B DNA maybe considered for participation, but must agree to receive appropriate anti-hepatitis B viral therapy suppression therapy while on obinutuzumab and have hepatitis B DNA monitored every 4 weeks with real-time polymerase chain reaction (PCR) by the treating physician; these patients should be referred to a hepatologist or gastroenterologist for appropriate monitoring and management
  * Hepatitis C: patients with positive hepatitis C serology unless hepatitis C virus (HCV) ribonucleic acid (RNA) is confirmed negative by PCR
* Vaccination with a live vaccine a minimum of 28 days prior to the start of treatment
* Patient is receiving other investigational drugs
* Prior chemotherapy for any other cancer within the last 2 years
* Patients should not have active or uncontrolled autoimmune hemolytic anemia or immune thrombocytopenia
* Patients should not have transfusion-dependent thrombocytopenia or bleeding disorders
* Patients should not have an autoimmune disorder that requires active immunosuppression
* Patients should not have a history of uncontrolled seizures
* Currently active, clinically significant cardiovascular disease, such as uncontrolled arrhythmia or class 3 or 4 congestive heart failure as defined by the New York Heart Association functional classification; or a history of myocardial infarction, unstable angina, or acute coronary syndrome within 6 months prior to enrollment on the study
* Patients should not have a stroke or intracranial hemorrhage within last 6 months
* Prior surgery: patients may not have had major surgery within 28 days of enrollment, or minor surgery within 7 days of enrollment; examples of minor surgery include dental surgery, insertion of a venous access device, skin biopsy, or aspiration of a joint; the decision about whether a surgery is major or minor can be made at the discretion of the treating physician
* Any life-threatening illness, medical condition, or organ system dysfunction that, in the investigator's opinion, could compromise the subject's safety or put the study outcomes at undue risk
* Pregnant and nursing: female patients must have a negative serum pregnancy test within 72 hours prior to initiating protocol therapy and be practicing an effective form of contraception during protocol therapy and for at least 4 weeks following completion of protocol therapy
* Currently active, clinically significant hepatic impairment Child-Pugh class B or C according to the Child Pugh classification

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2018-02-20 (Actual); Primary Completion 2026-09-11 (Estimated); Study Completion 2032-02-20 (Estimated)

PRIMARY OUTCOMES:
Overall response rate in patients with newly diagnosed indolent lymphoma requiring treatment, including complete response and partial response | Two years
  Response will be assessed by the revised Lugano. Will compute estimates of response, along with corresponding confidence intervals, using appropriate exact methods that take into account the 2-stage design.

SECONDARY OUTCOMES:
Partial remission or complete remission in patients treated with ibrutinib and obinutuzumab | Two years
  Response will be assessed by the revised Lugano. Will compute estimates of response, along with corresponding confidence intervals, using appropriate exact methods that take into account the 2-stage design.
Progression free survival | 1 year
  Estimated using Kaplan-Meier method.
Progression free survival | 3 years
  Estimated using Kaplan-Meier method.
Progression free survival | 5 years
  Estimated using Kaplan-Meier method.
Overall survival | 1 year
  Estimated using Kaplan-Meier method.
Overall survival | 3 years
  Estimated using Kaplan-Meier method.
Overall survival | 5 years
  Estimated using Kaplan-Meier method.
Incidence of grade III-IV toxicity | Two years
  Assessed using Common Terminology Criteria for Adverse Events version 5.0. Will compute estimates toxicity rates, along with corresponding confidence intervals, using appropriate exact methods that take into account the 2-stage design.

CONTACTS AND LOCATIONS:
Overall Officials: Ubaldo Martinez-Outschoorn, MD, Principal Investigator — Sidney Kimmel Cancer Center at Thomas Jefferson University
Locations (1):
- Sidney Kimmel Cancer Center at Thomas Jefferson University, Philadelphia, Pennsylvania, United States

REFERENCES:
- See also: Thomas Jefferson University Hospital — http://hospitals.jefferson.edu/